CLINICAL TRIAL: NCT03539159
Title: Allogenic Serum Micro Eye Drops Compared to Conventional Sized Eye Drops: A Prospective Randomized Non-inferiority, Investigator Masked, Cross-over Multicenter Clinical Study
Brief Title: Assessment of the Mu-Drop System for Serum Eye Drops
Acronym: AmuSED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Radboud University Medical Center (Other); Leiden University Medical Center (Other); UMC Utrecht (Other); Maastricht University Medical Center (Other); Amsterdam UMC, location AMC (Other); The Rotterdam Eye Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL63119.091.17
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Dry Eye Syndrome
Keywords: Allogeneic serum eye drops; Micro eye drops; Cross-over multicenter trial; Ocular Surface Disease Index (OSDI)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic conventional sized serum eye drops (Experimental)
  Interventions: Other: Allogeneic conventional sized serum eye drops; Other: Allogeneic micro sized serum eye drops
- Allogeneic micro sized serum eye drops (Experimental)
  Interventions: Other: Allogeneic conventional sized serum eye drops; Other: Allogeneic micro sized serum eye drops

INTERVENTIONS:
Other: Allogeneic conventional sized serum eye drops — allogeneic serum conventional sized drops (40-50 µL, administrated using the Meise applicator) applied six times a day (when appropriate, lowering the dose to 3-4 times a day is allowed) for a period of one month
Other: Allogeneic micro sized serum eye drops — Allogeneic serum micro eye drops (5-10 µL, administrated using the mu-Drop applicator) applied six times a day (when appropriate, lowering the dose to 3-4 times a day is allowed) for a period of one month

SUMMARY:
Rationale: Serum eye drops (SEDs) are used to treat patients with severe signs and symptoms of dry eyes and other corneal defects. Serum is used in severe ophthalmic cases where conventional treatment and/or eye drops (artificial tears) have insufficient effect. The use of SEDs in dry eye patients usually has a rapid effect. Most patients claim the effect to be instantaneous, and most symptoms improve within 48-72 hours.

There is evidence suggesting that substances in serum may help in the healing of epithelial defects, such as epidermal growth factor, fibroblast growth factor, fibronectin, and/or vitamin A. However, the precise serum factor responsible for alleviating the patient's complaints is currently not known.

SEDs are considered as a blood product under EU blood legislation (Directive 2002/98/EC), as well as in New Zealand and Australia. Commonly, autologous SEDs are used, but they are replaced more and more by allogeneic SEDs prepared from donor serum. Allogeneic SEDs are derived from healthy voluntary, non-remunerated male donors with blood group AB, and have the benefit of blood bank controlled quality. They can be delivered from stock and are therefore quickly available for each patient.

For application of eye drops, generally administration systems with a drop size of 40 to 50 µl are used, further on referred to as conventional sized eye drops. From previous studies done with medicinal eye drops, it has been shown that smaller eye drops, so called micro drops, can be just as effective and sometimes even superior to conventional drops for treatment of eye disease. If micro drops are just as effective or maybe even superior to conventional sized eye drops is currently unknown for the use of SEDs. This study will compare the feasibility and effectiveness of allogeneic serum micro eye drops using the mu-Drop applicator to the conventional sized allogeneic eye drops using the Meise applicator. Both systems have a closed manufacturing system.

Objective: The main objective is to determine whether the administration of allogeneic serum micro eye drops is non-inferior in terms of effectiveness and safety as compared to the conventional sized drops.

Main study parameters/endpoints: The primary endpoint is the improvement in OSDI score by using SEDs (OSDI score after treatment minus OSDI score before treatment), independent of the drop size, showing non-inferiority for the use of micro drops as compared to conventional sized drops.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe signs and symptoms of dry eyes.
* Age 16 years or older.
* Punctate staining of the cornea.
* Expected to benefit from SEDs.
* Not previously treated with SEDs.

Exclusion Criteria:

* Actively or previously treated for Herpes Simplex Virus (HSV) keratitis.
* Corneal lesions, more than punctate.
* Untreated Meibomian gland disease.
* Pregnant or lactating or intending to become pregnant in the next 3 months
* Unable or unwilling to give informed consent.
* Active (systemic) microbial infection.
* The use of all types of contact lenses.
* Discontinuous use of medication that affects the dry eye sensation is not allowed (e.g. discontinuous use of local corticosteroids). Continuous use of co-medication, like lubricants, anti-glaucoma eye drops or other drops, that have to be used on a daily basis are allowed, and are expected to be used throughout the study period in both eyes (continuous use of the same medication is allowed if used at least one month prior to start of the study).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI index) | One month after starting the intervention
  The primary endpoint is the improvement in OSDI score by using SEDs (OSDI score after treatment minus OSDI score before treatment), independent of the drop size, showing non-inferiority for the use of micro drops as compared to conventional sized drops. The OSDI score falls between 0 and 100, ranging from normal, mild, moderate to severe dry eyes.

SECONDARY OUTCOMES:
Schirmer's test | One month after starting the intervention
  Tear production in mm
Tear break up time | One month after starting the intervention
  number of seconds the dry spot appears in the ter film
Corneal punctates | One month after starting the intervention
  Percentage of affected surface after staining of the cornea

CONTACTS AND LOCATIONS:
Overall Officials: Cathrien Eggink, MD, Principal Investigator — Radboud University Medical Center
Locations (6):
- Netherlands (6):
  - Academic Medical Center Amsterdam, Amsterdam-Zuidoost
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboudumc, Nijmegen
  - The Rotterdam Eye Hospital, Rotterdam
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Vermeulen C, van der Burg LLJ, van Geloven N, Eggink CA, Cheng YYY, Nuijts RMMA, Wisse RPL, van Luijk CM, Nieuwendaal C, Remeijer L, van der Meer PF, de Korte D, Klei TRL. Allogeneic Serum Eye Drops: A Randomized Clinical Trial to Evaluate the Clinical Effectiveness of Two Drop Sizes. Ophthalmol Ther. 2023 Dec;12(6):3347-3359. doi: 10.1007/s40123-023-00827-5. Epub 2023 Oct 16. PMID 37843772